CLINICAL TRIAL: NCT04807881
Title: An Exploratory Clinical Study of Keynatinib in Relapsed/Refractory B-cell Lymphoma
Brief Title: Phase Ib Clinical Study of Keynatinib
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medolution Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDO-BTK-20001
Record Dates: First submitted 2021-03-18; First posted 2021-03-19 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Lymphoma, B-Cell
Keywords: Relapsed/Refractory Primary Central Nervous System Lymphoma; Relapsed/Refractory Chronic Lymphoblastic Leukemia; Relapsed/Refractory Small Lymphocytic Lymphoma; Relapsed/Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Keynatinib treatment group (Experimental): Keynatinib, 20 mg，BID
  Interventions: Drug: Keynatinib

INTERVENTIONS:
Drug: Keynatinib — All subjects shall be treated with Keynatinib twice a day (once every 12 hours), 20 mg each time, fasting within 2 hours before and 1 hour after taking the drug, and taking warm water when taking the drug. It is recommended to take the drug at the same time every day. In case of missed administration, the subjects should be instructed to take it as soon as possible when they think of it on the same day. If it is within 3 hours later than the scheduled administration, the study drug should be taken as soon as possible; if the interval is > 3 hours, skip this time and take the next dose at the normal scheduled time. Do not take double dose at one time. Every 28 days is a treatment cycle until the specified interview completed, PD, intolerable toxicity, death occurs or withdraw from the study (including withdrawal of informed consent by the subject or termination of the study when the investigator judges that the risk is greater than the benefit), whichever occurs first.
  Other Names: TL007

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, PK characteristics in subjects with relapsed/refractory B-cell lymphoma. Furthermore, the relationship between the exposure level of Keynatinib and its efficacy and safety, the penetration rate of keynatinib in the Blood-Brain Barrier (BBB) and its PK characteristics in cerebrospinal fluid in R/R-PCNSL patients, the relationship between the BTK receptor occupancy rate and the efficacy are also evaluated.

DETAILED DESCRIPTION:
This tiral adopts a multi-center, single-arm, multi-cohort, and open-label design to evaluate the efficacy and safety of keynatinib in patients with relapsed/refractory B-cell lymphoma.

There will be three cohorts in this trial, details as follows: Cohort 1: R/R-PCNSL subjects; Cohort 2: R/R-CLL/SLL subjects; Cohort 3: R/R-MCL subjects.

10-25 subjects will be enrolled in the R/R-PCNSL, R/R-CLL/SLL, and R/R-MCL cohorts, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Unlimited gender, age ≥ 18 years (including critical value)-Cohort 1/2/3;
2. Voluntarily participate in the study and sign the ICF, follow the trial treatment protocol and interview plan-Cohort 1/2/3;
3. The subject's disease diagnosis meets all of the following conditions:

   Cohort 1:
   1. Primary central nervous system lymphoma (PCNSL) confirmed by pathology;
   2. For relapsed or refractory PCNSL, at least first line treatment must be given to Central Nervous System (CNS) lesions;
   3. Brain Magnatic resonance Imaging (MRI) or Computerized tomography (CT) shows solid lesions of PD;

   Cohort 2:
   1. CLL/SLL diagnosed according to IWCLL 2008 standards;
   2. Refractory or relapsed CLL/SLL that previously received at least first-line systemic treatment. First-line treatment is defined as at least 2 cycles of standard protocol or clinical trial research protocol completed based on current guidelines;
   3. Accord with at least one indication of CLL / SLL that requiring treatment;
   4. There is medical record confirming that it is invalid or Progression Disease occurs after response for the latest treatment;
   5. CT /MRI shows measurable lesions, which is defined as at least one lymph node with a maximum axis of more than 1.5 cm and with 2 measurable vertical dimension;
   6. It is allowed to include the patients with a stable condition involving the central nervous system;

   Cohort 3:
   1. Mantle cell lymphoma diagnosed by histopathology: including that t (11; 14) (q13; q32) positive by cytogenetic test and / or cyclin D1 highly expressed by immunohistochemistry;
   2. Who have been pretreated with > 1 but failed in ≤ 3 different chemotherapies and / or targeted drugs treatment.
   3. There is a medical record confirming that it is invalid or Progression Disease occurs after response for the latest treatment;
   4. CT / MRI shows measurable lesions, which is defined as the longest diameter (of ≥1 lymph node) > 1.5 cm, and 2 vertical diameters is clearly measurable;
   5. It is allowed to include the patients with a stable condition involving the central nervous system;
4. When screening, the status score of Eastern Cooperative Oncology Group (ECOG) is 0 to 2 points-Cohort 1/2/3;
5. Estimated survival time ≥ 4 months-Cohort 1/2/3;
6. Subjects have appropriate organ functions, the main organ functions meet the following criteria:

   1. Blood routine: Neutrophil absolute value ≥ 1.0(in cohort1, 0.75 in cohort 2/3)×109 /L, platelet ≥ 75(in cohort1, 50 in cohort 2/3, 30×109/L are acceptable if CLL patients have bone marrow involvement, transfusion-dependent thrombocytopenia is excluded )×109 /L, hemoglobin ≥ 80 g/L(in cohort1). [No blood transfusion and hematopoietic stimulating factor are used within 21 days (7 days in cohort 2/3) before the first administration-Chort1];
   2. Blood biochemistry: Total bilirubin (TBIL) ≤ 2 × ULN (unless diagnosed as Gilbert syndrome), Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 × ULN; serum creatinine ≤ 2 × ULN or creatinine clearance rate ≥ 50 ml / min (calculated according to Cockcroft Gault formula)-Cohort 1/2/3;
   3. Coagulation function: International Standardized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN-Cohort 1/2/3;
7. Fertile female subjects must agree to use contraceptives with an annual failure rate of < 1% or maintain abstinence (avoid heterosexual intercourse) during the study and at least 90 days after the last administration of the study drug. Contraceptive methods with an annual failure rate of <1% includes bilateral tubal ligation, male sterilization, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing IUD (intrauterine devices), and copper-containing IUD. Male subjects must be sterilized by vasectomy or barrier contraception, and female partners should use the effective contraceptives as described above. In addition, male subjects are not allowed to donate sperm within 90 days after the last administration-Cohort 1/2/3.

Exclusion Criteria:

* Cohort 1: R/R-PCNSL

  1. PCNSL is pathologically diagnosed as T-cell lymphoma;
  2. Have previously received any of the following treatments:

     1. Chemotherapy, targeted therapy, radiotherapy or antibody based anti-tumor therapy are used within 4 weeks before the first administration or within 5 half-lives (whichever is shorter);
     2. Have previously received the treatment of B Cell Receptor (BCR) inhibitors (such as BTK, phosphoinositide kinase 3 kinase [PI3K] or SYK inhibitors) or BCL-2 inhibitors (such as ABT-199) or Chimeric Antigen Receptor T-Cell Immunotherapy (CAR-T) or a bispecific antibody drug;
     3. Have received Allogenetic Haematopoietic Stem Cell Transplantation (Allo-HSCT) or other organ transplants (except for those who have received ASCT more than six months);
  3. Take ≥ 8 mg dexamethasone or equivalent daily to control lymphoma symptoms;
  4. CNS external beam radiotherapy within 21 days before the first administration;
  5. The systemic immunosuppressants, including cyclosporine A, tacrolimus, sirolimus and other drugs, haven't stopped 28 days before the first use of the study drug, or > 5 mg/day of prednisone or its equivalent has been taken for long period;
  6. Have other malignant tumors within 3 years, except for the curable basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of cervix or breast;
  7. Non-hematologic toxicity of the previous anti-tumor treatment has not recovered to ≤ grade 1 (except for hair loss);
  8. Have uncontrollable or severe cardiovascular disease, including:

     1. Congestive heart failure with New York Heart Association (NYHA) grade II or higher, unstable angina, myocardial infarction within 6 months before first study drug administration, or arrhythmia requiring treatment during screening, Left Ventricular Ejection Fraction (LVEF) <50% ;
     2. Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, and atypical cardiomyopathy);
     3. Clinically significant QTc interval prolonged medical history, or the QTc interval of screening period > 470 ms in female, and > 450 ms in male;
     4. Uncontrollable high blood pressure (on the basis of improving life style, with 2 or more antihypertensive drugs (including diuretics) that will be reasonably tolerable and sufficient for more than one month being applied, the blood pressure has not reached to the standard yet, or the blood pressure could only be effectively controlled by taking 4 or more antihypertensive drugs);
  9. Have active bleeding within 2 months before screening or are taking anticoagulant/antiplatelet drugs, or the investigators believe that there is a clear bleeding tendency (such as esophageal varices with bleeding risk, or a locally active ulcer lesions);
  10. Have medical history of deep vein thrombosis or pulmonary embolism;
  11. Have medical history of stroke or intracranial hemorrhage within 6 months before taking the study drug, except for intracranial hemorrhage due to surgical sequelae;
  12. Have clinically significant gastrointestinal abnormalities, which might affect drug intake, transport or absorption (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
  13. Have serious or active infection requiring systematic anti infection treatment;
  14. At screening, patients with active uncontrolled infection [such as infection that requiring intravenous antibiotic therapy, human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, etc.]; Note: If hepatitis B virus surface antigen (HBsAg) is positive, HBV-DNA < 1000 cop/ml, and ALT/AST ≤ 2.0 × ULN can be included. HCV infection is defined as HCV-Ab positive.
  15. Have past history of or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc;
  16. Have undergone major surgery or have not recovered from the invasive operation within 4 weeks before taking the study drug for the first time and are not suitable for the clinical trial according to the judgment of the investigators;
  17. Who is participating in other clinical studies or have participated in other intervention clinical trials within 4 weeks before screening;
  18. Have history of alcohol or drug abuse;
  19. Pregnant or lactating women;
  20. Concomitant administration of drugs with moderate to severe inhibition or strong induction of cytochrome P450 CYP3A
  21. Subjects determined by the investigators to be unsuitable for other reasons;

Cohort 2: R/R-CLL/SLL

1. Have medical history of prolymphocytic leukemia, known medical history of Richter syndrome or currently suspected Richter transformation (patients with clinical suspicion need biopsy to exclude transformation)
2. Have previously received any of the following treatments:

   1. Chemotherapy, targeted therapy, radiotherapy or antibody-based anti-tumor therapy within 4 weeks or 5 half-lives (whichever is shorter) before the first administration;
   2. Previous treatment with BTK, phosphoinositide kinase 3 kinase [PI3K] or SYK inhibitors or BCL-2 inhibitors (such as ABT-199) or chimeric antigen receptor T cell immunotherapy (CAR-T) or treatment with bispecific antibody drugs;
   3. Patients who received allogeneic hematopoietic stem cell transplantation (Allo-HSCT) or other organ transplantation within the past 6 months;
   4. Patients who received autologous hematopoietic stem cell transplantation within the past 6 months;
3. Use of systemic corticosteroids within 7 days before the first administration of study drug, or continuous use of prednisone at or above 20 mg/day or equivalent;
4. Other malignancies within 3 years, except for curable basal or squamous cell skin cancer, superficial bladder cancer, and carcinoma in situ of the uterine cervix or breast;
5. Non-hematologic toxicity of the previous anti-tumor treatment has not recovered to ≤ grade 1 (except for hair loss);
6. Have uncontrollable or severe cardiovascular disease, including:

   1. Congestive heart failure with New York Heart Association (NYHA) grade II or higher, unstable angina, myocardial infarction within 6 months before first study drug administration, or arrhythmia requiring treatment during screening period, Left Ventricular Ejection Fraction (LVEF) <50%;
   2. Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, and atypical cardiomyopathy);
   3. Clinically significant QTc interval prolonged medical history, or the QTc interval of screening period > 470 ms in female, and > 450 ms in male;
   4. Uncontrollable high blood pressure (on the basis of improving life style, with 2 or more antihypertensive drugs (including diuretics) being applied that will be reasonably tolerable and sufficient for more than one month, the blood pressure has not reached to the standard yet, , or the blood pressure could only be effectively controlled by taking 4 or more antihypertensive drugs);
7. Have active bleeding within 2 months before screening or is taking anticoagulant/antiplatelet drugs, or the investigators believe that there is a clear bleeding tendency (such as esophageal varices with bleeding risk, or a locally active ulcer lesions);
8. Active and/or persistent autoimmune anemia and/or autoimmune thrombocytopenia requiring treatment (e.g., idiopathic thrombocytopenic purpura);
9. Have medical history of deep vein thrombosis or pulmonary embolism;
10. Have medical history of stroke or intracranial hemorrhage within 6 months before taking study drug;
11. Have clinically significant gastrointestinal abnormalities, which might affect drug intake, transport or absorption (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
12. Have active infection requiring systemic anti-infective treatment;
13. At screening, patients with active uncontrolled infection [such as intravenous infection that requiring antibiotic therapy, human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, etc.]; Note: If hepatitis B virus surface antigen (HBsAg) is positive, HBV-DNA < 1000 cop/ml, and ALT/AST ≤ 2.0 × ULN can be included. HCV infection is defined as HCV-Ab positive.
14. Have past history of or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc;
15. Have history of alcohol or drug abuse;
16. Have undergone major surgery or have not recovered from the invasive operation within 4 weeks before taking the study drug for the first time and are not suitable for the clinical trial according to the judgment of the investigators;
17. Whowill participating in other clinical studies or haveparticipated in other intervention clinical trials within 4 weeks before screening;
18. Pregnant or lactating women;
19. Concomitant administration of drugs with moderate to severe inhibition or strong induction of cytochrome P450 CYP3A;
20. Subjects determined by the investigators to be unsuitable for other reasons;

Cohort 3: R/R-MCL

1. Havepreviously received any of the following treatments:

   1. Chemotherapy, targeted therapy, radiotherapy or antibody based anti-tumor therapy are used within the first 4 weeks or 5 half-lives (whichever is shorter) before the first administration;
   2. Have previously received the treatment of BTK, phosphoinositide kinase 3 kinase [PI3K] or SYK inhibitors) or BCL-2 inhibitors (such as ABT-199) or Chimeric Antigen Receptor T-Cell Immunotherapy (CAR-T) or received bispecific antibody drug;
2. Use of systemic corticosteroids at or above 20 mg/day prednisone or equivalent within 7 days before the first administration of study drug;
3. Have other malignant tumors within 3 years, except for the curable basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of cervix or breast ;
4. Non-hematologic toxicity of the previous anti-tumor treatment has not recovered to ≤ grade 1 (except for hair loss);
5. Have uncontrollable or severe cardiovascular disease, including:

   1. Congestive heart failure with New York Heart Association (NYHA) grade II or higher, unstable angina, myocardial infarction within 6 months before first study drug administration, or arrhythmia requiring treatment during screening period, Left Ventricular Ejection Fraction (LVEF) <50% ;
   2. Primary cardiomyopathy (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, and atypical cardiomyopathy);
   3. Clinically significant QTc interval prolonged medical history, or the QTc interval of screening period > 470 ms in female, and > 450 ms in male;
   4. Uncontrollable high blood pressure (on the basis of improving life style, with 2 or more antihypertensive drugs (including diuretics) that will be reasonably tolerable and sufficient for more than one month being applied, the blood pressure has not reached to the standard yet, , or the blood pressure could only be effectively controlled by taking 4 or more antihypertensive drugs);
6. Have medical history of deep vein thrombosis or pulmonary embolism;
7. Have medical history of stroke or intracranial hemorrhage within 6 months before taking study drug;
8. Have clinically significant gastrointestinal abnormalities, which might affect drug intake, transport or absorption (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
9. Have serious or active infection requiring systematic anti infection treatment;
10. At screening, patients with active uncontrolled infection [such as infection that requiring intravenous antibiotic therapy, human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, etc.]; Note: If hepatitis B virus surface antigen (HBsAg) is positive, HBV-DNA < 1000 cop/ml, and ALT/AST≤ 2.0 × ULN can be included. HCV infection is defined as HCV-Ab positive.
11. Have past history of or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc;
12. Have history of alcohol or drug abuse;
13. Have undergone major surgery or have not recovered from the invasive operation within 4 weeks before taking the study drug for the first time and is not suitable for the clinical trial according to the judgment of the investigators;
14. Who is participating in other clinical studies or have participated in other intervention clinical trials within 4 weeks before screening;
15. Pregnant or lactating women;
16. Concomitant administration of drugs with moderate to severe inhibition or strong induction of cytochrome P450 CYP3A;
17. Subjects determined by the investigators to be unsuitable for other reasons;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2027-10-10 (Estimated); Study Completion 2028-04-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (CR+PR) | Every 2 administration cycles in cycle 1-6 and every 3 administration cycles in cycle 7-n.
  The proportion of subjects whose optimal efficacy observed from the beginning of administration is CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: Dawei Zhang, phD, Study Director — Medolution Ltd.
Locations (4):
- China (4):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.